CLINICAL TRIAL: NCT05552664
Title: The Genetic Information and Family Testing (GIFT) Study
Acronym: GIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: UMCC 2022.066; HUM00224851 (Other: University of Michigan); U01CA254822 (NIH); HUM00221150 (Other: University of Michigan)
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Genetic Testing; Family testing
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial is a 2x2 factorial prospective RCT
Who Masked: Participant
Masking Description: Randomization will be concealed from study participants; enrolled patients and relatives will not be aware that their family has been randomized into one of four trial arms and provided a different intervention experience than the other study participants. Concealment is necessary for this study so that the trial can observe differences across the trial arms without a) negatively impacting study enrollment and biasing the study, and b) causing unnecessary negative emotional reactions in study participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Other): Arm information details will not be provided at this time in order to preserve scientific integrity and will be updated once the study has resulted.
  Interventions: Genetic: GIFT
- Arm 2 (Other): Arm information details will not be provided at this time in order to preserve scientific integrity and will be updated once the study has resulted.
  Interventions: Genetic: GIFT
- Arm 3 (Other): Arm information details will not be provided at this time in order to preserve scientific integrity and will be updated once the study has resulted.
  Interventions: Genetic: GIFT
- Arm 4 (Other): Arm information details will not be provided at this time in order to preserve scientific integrity and will be updated once the study has resulted.
  Interventions: Genetic: GIFT

INTERVENTIONS:
Genetic: GIFT — GIFT features a web-based intervention that offers access to an online family communication program containing key facts about genetics, cancer risk, and the role of genetic testing and helps patients share health information with their first-and second-degree relatives, whom they can invite to join the study to receive education/support and access to low-cost genetic testing.

SUMMARY:
The Genetic Information and Family Testing (GIFT) Study is designed to support the capacity, opportunity, and motivation of cancer patients to engage their relatives about inherited cancer susceptibility and provide support and services to those relatives to initiate GRE (including genetic testing) and prepare them to subsequently engage their clinicians in informed decision-making about cancer prevention and early detection.

DETAILED DESCRIPTION:
GIFT features a web-based intervention that offers access to an online family communication program containing key facts about genetics, cancer risk, and the role of genetic testing and helps patients share health information with their first-and second-degree relatives, whom they can invite to join the study to receive education/support and access to low-cost genetic testing. Two design features of the intervention will be randomized and evaluated to determine the best approach for future scalability.

Those eligible will be offered enrollment into the Michigan-hosted intervention trial, and those who enroll will be randomized into 1 of 4 study arms. Patients can invite their relatives to enroll and receive genetic testing via Color. Families randomized to the arms with human Navigator support will also have access to a Family Health Navigator at Stanford University. Enrolled patients and relatives will be surveyed six months post-enrollment to collect additional information regarding their interactions with the GIFT platform and their experiences with genetic risk evaluation.

Study phase and approximate sample size is summarized below:

* Initial patient sample selected- 5250 patients
* Respondents to PICS survey- 3150 patients
* Pool of patients eligible for GIFT study invitation- 2930 patients
* Patient GIFT study participants- 880 patients
* Relatives invited to the GIFT study- 3520 relatives
* Relative GIFT study participants- 1584 relatives

Study phase and approximate sample size summarizes have been updated below and IRB approved 29SEP2025:

* Initial patient sample selected- 4300 patients
* Respondents to PICS survey- 2358 patients
* Pool of patients eligible for GIFT study invitation- 2030 patients
* Patient GIFT study participants- 412 patients
* Relatives invited to the GIFT study- 1236 relatives
* Relative GIFT study participants- 371 relatives

ELIGIBILITY:
Inclusion criteria for the PICS survey are:

1. diagnosed with any cancer at any stage in 2018-2019 and reported to the Georgia or California SEER registries
2. Been found to carry a pathogenic variant (PV) in one of 27 cancer susceptibility genes (see Table 4) according to the Georgia California Genetic Testing Linkage Initiative dataset
3. aged 18 or older
4. alive at the time of selection as determined through linkage with Georgia and California vital statistics data.

Additional eligibility criteria for Patient Trial Invitation will be evaluated from patient response to the PICS survey and will include patient report of:

1. Receipt of genetic testing for cancer risk
2. A positive test result (pathogenic variant; PV)

Inclusion criteria for Relative Trial Invitation are assessed via patient report:

1. first-degree (biological parent, sibling, or biological child) or second-degree (biological half-sibling, aunt, uncle, nephew, niece, grandparent, or grandchild) relative of a patient enrolled in the study;
2. aged 18 or older;
3. alive at the time of study invitation;
4. relative lives in the United States or Canada (countries in which Color genetic testing is available, most people speak either English or Spanish, and test kit shipping costs are not exorbitant)

Additional eligibility criteria for Relative Trial Enrollment will be evaluated from relative response to the relative eligibility screening survey (see Appendix C) and will include:

1. confirmation from the relative that they have not received clinical genetic testing ordered by a doctor or genetic counselor within the past five years (proxy for having already been tested for the PV carried by the patient who invited them into the study);
2. confirmation of age 18 or older;
3. confirmation of first-degree (biological parent, sibling, or biological child) or second-degree (biological half-sibling, aunt, uncle, nephew, niece, grandparent, or grandchild) relation to the patient.
4. confirmation of residence in United States or Canada

Exclusion Criteria

Exclusion criteria for the PICS survey are:

1) Age<18

Additional exclusion criteria for Patient Trial Invitation:

1. Patients who do not report receipt of genetic testing
2. Patients who do not report a positive genetic test result (PV)

Exclusion criteria for Relative Trial Invitation are:

1. Age<18
2. Relative does not live in the United States or Canada

Additional exclusion criteria for Relative Trial Enrollment include relative report of:

1. Age<18;
2. Receipt of genetic testing ordered by a doctor or genetic counselor within the past five years;
3. Relationship to proband (inviting) patient other than first- or second-degree relative
4. Residence in a country other than United States or Canada

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3002 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
To determine the independent effects of the two virtual platform design features on relatives' receipt of genetic testing. | 6 months after the final relative enrolls
  The proportion of each enrolled patient's 1st and 2nd degree relatives who receive Color genetic testing through the GIFT platform.
  For each enrolled patient, this will be calculated as the number of enrolled relatives who obtain a genetic test result from Color (complete the genetic testing process) via the GIFT Study divided by the number of relatives reported on the baseline PICS survey. The endpoint of interest is the presence (as opposed to the absence) of a test result (e.g., positive, uncertain, negative) on the Color Quarterly Report.
  Assessed six months after the final relative enrolls in the study.

SECONDARY OUTCOMES:
To determine the independent effects of the two virtual platform design features on the proportion of relatives invited by each patient to enroll in the study. | 91 days after the final patient enrolls
  The proportion of each enrolled patient's relatives who are invited to join the study. For each enrolled patient:
  Number of invited relatives / Number of relatives reported on baseline PICS survey
  Assessed 91 days after the final patient enrolls in the study.
To determine the independent effects of the two virtual platform design features on the cancer patients' assessment of communication with their relatives about hereditary cancer and genetic risk evaluation. | After the 6 month follow up survey
  A 20-item scale with responses on a 5-point Likert from "not at all true" to "very true." Items assess patients' capacity, opportunity, and motivation to communicate with family members about their genetic test results. The outcome is continuous and we will measure the change in mean score from baseline to follow-up survey. A greater difference between timepoints will indicate greater improvement in the patient's assessment of their communication with relatives.
  Assessed at two time points: baseline PICS survey and Patient Six-Month Follow-up Survey.
To determine the independent effects of the two virtual platform design features on relatives' receipt of a formal cancer genetic counseling session in practice. | After the 6 month follow up survey
  Single question on a binary yes/no scale. Yes will indicate receipt of formal GRE.
  Assessed in the Relative Six-Month Follow-Up Survey

CONTACTS AND LOCATIONS:
Overall Officials: Steven Katz, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan

REFERENCES:
- [Derived] Katz SJ, Abrahamse P, Hofer TP, Courser RR, Hodan R, Tocco RS, Rios-Ventura S, Ward KC, Hamilton AS, Kurian AW, An LC. The Genetic Information and Family Testing (GIFT) study: trial design and protocol. BMC Cancer. 2025 Feb 27;25(1):366. doi: 10.1186/s12885-025-13744-6. PMID 40016666